CLINICAL TRIAL: NCT01299987
Title: TARGIT-E(Elderly) Prospective Phase II Study of Intraoperative Radiotherapy (IORT) in Elderly Patients with Small Breast Cancer
Brief Title: Prospective Phase II Study of Intraoperative Radiotherapy (IORT) in Elderly Patients with Small Breast Cancer
Acronym: TARGIT-E
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsmedizin Mannheim (Other)
Responsible Party: Principal Investigator, Elena Sperk, MD, Managing Director Mannheim Cancer Center Clinical Trials Unit, Heidelberg University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TARGIT-E
Record Dates: First submitted 2011-02-18; First posted 2011-02-21 (Estimated); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Breast Neoplasms; Breast Diseases; Neoplasm Recurrence, Local; Neoplasms
Keywords: Keywords provided by University Hospital Mannheim:; Intraoperative Radiotherapy; Early Breast Cancer; Elderly Patients
MeSH Terms: conditions — Breast Neoplasms; Breast Diseases; Neoplasm Recurrence, Local; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intraoperative radiotherapy (Experimental): single arm with intraoperative radiotherapy
  Interventions: Radiation: intraoperative radiotherapy

INTERVENTIONS:
Radiation: intraoperative radiotherapy — intraoperative single dose radiotherapy (20 Gy)
  Other Names: IORT

SUMMARY:
This prospective, multicentric single arm phase II study is based on the protocol of the international TARGIT-A study. The purpose is to investigate the efficacy of a single intraoperative radiotherapy treatment within elderly low risk patients (≥ 70 years, cT1, cN0, cM0, invasive-ductal) which is followed by WBRT only when risk factors are present. In presence of risk factors postoperative WBRT will be added to complete the radiotherapeutic treatment according to international guidelines.

DETAILED DESCRIPTION:
Patients ≥ 70 years with small, low-risk breast cancer who are operated but not irradiated show local relapse rates around 4% after 4 years. With adjuvant whole breast radiotherapy (WBRT) the local relapse rate drops to 1% after 4 years under Tamoxifen (Hughes et al 2004). It has been demonstrated (Polgar et al. 2007, Vaidya et al. 2010) that the efficacy of radiation of the tumor bed only in a selected group can be non-inferior to WBRT. The TARGIT E study should confirm the efficacy of a single dose of intraoperative radiotherapy (IORT) in a well selected group of elderly patients with small breast cancer and absence of risk factors. In presence of risk factors postoperative WBRT will be added to complete the radiotherapeutic treatment according to international guidelines.

Endpoints are the local relapse rate (within 2 cm of the tumor bed), ipsilateral relapse, cancer-specific and overall survival and contralateral breast cancer as well as documentation of quality of life and cosmetic outcome. The expected local relapse rates are 0.5/1/1.5% after 2.5/5/7.5 years, respectively.

Discontinuation of the trial is scheduled if rates of local relapse rates rise to 3/4/6% after 2.5/5/7.5 years. Power calculations result in 265 patients with a calculated loss to follow-up of 20%, an alpha of 0.05 and a beta 0.1. Only centers with access to the Intrabeam® system (Carl Zeiss) can recruit patients into the trial.

ELIGIBILITY:
Inclusion Criteria:

* cT1c cN0 cM0
* ≥ 70 years old
* invasive-ductal histology
* compliance
* informed consent

Exclusion Criteria:

* extensive intraductal component (EIC)
* multifocality /-centricity
* lymph vessel invasion (L1)
* clinical signs of distant metastases or clinically suspicious lymph nodes
* other histology
* < 70 years old
* missing informed consent or non-compliance
* bilateral breast cancer at time of diagnosis
* known BRACA 1/2 mutations (genetic testing not required)

Min Age: 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 591 (Actual)
Dates: Start 2011-01 (Actual); Primary Completion 2022-11 (Actual); Study Completion 2022-11 (Actual)

PRIMARY OUTCOMES:
Local Relapse | up to ten years
  Rate of local relapse (within 2cm of the initial tumor bed)

SECONDARY OUTCOMES:
Overall Survival | up to ten years
  Death is an event
Ipsi- or Contralateral Breast Cancer | up to ten years
  Rate of ipsilateral and contralateral breast cancer events
Cosmesis | up to 7.5 years
  BCCT.Core analysis of cosmesis
General and breast-specific Quality of Life after IORT | up to 10 years
  EORTC questionnaires QLQ C30 and BR23
Late toxicity after IORT | up to ten years
  LENT-SOMA based toxicity at all FU time points

CONTACTS AND LOCATIONS:
Overall Officials: Sperk Elena, MD, Principal Investigator — Medical Faculty Mannheim
Locations (1):
- Universitätsmedizin Mannheim UMM, Mannheim, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: No
It was not planned initially back in 2011.

REFERENCES:
- [Derived] Sperk E, Lemanski C, Neumaier C, Lauer J, Siefert V, Volker R, Lindner C, Niehoff P, Tallet AR, Racadot S, Petit A, Pazos M, Le-Blanc Onfroy M, Martin E, Reuter C, Hermann RM, Pohl F, Friedrichs K, Wurschmidt F, Pigorsch S, Kolberg HC, Graf H, Brunner TB, Malter W, Park-Simon TW, Brucker C, Fleckenstein J, Petersen C, Tuschy B, Wilken EE, Buttner S, Sutterlin M, Flyger H, Wenz F. Intraoperative radiotherapy in elderly patients with breast cancer: long-term follow-up results of the prospective phase II trial TARGIT-E. BMC Cancer. 2025 Dec 4;25(1):1862. doi: 10.1186/s12885-025-15289-0. PMID 41345599
- [Derived] Neumaier C, Elena S, Grit W, Yasser AM, Uta KT, Anke K, Axel G, Marc S, Frederik W. TARGIT-E(lderly)--prospective phase II study of intraoperative radiotherapy (IORT) in elderly patients with small breast cancer. BMC Cancer. 2012 May 8;12:171. doi: 10.1186/1471-2407-12-171. PMID 22569123